CLINICAL TRIAL: NCT04669353
Title: The Effect of Autologous Application of Platelet Rich Plasma on Wound Healing and Pain Perception After Cesarean Section in a Low Resource Setting
Brief Title: Platelet Rich Plasma and Wound Healing After Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Nabih Elkhouly, associate professor, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 198190PSGN33
Record Dates: First submitted 2020-12-06; First posted 2020-12-16 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Infection
Keywords: Platelet Rich Plasma; wound Healing; Pain; Cesarean Section
MeSH Terms: conditions — Infections; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The invesigators randomized participants in a 1:1 ratio to two equal groups containing one hundred patients each (intervention and control groups). A statistician not directly involved in the study prepared a computer generated randomization list and placed the allocation information in sequentially numbered sealed envelopes that were opened according to the attendance of the patients after signing the informed consent. The study authors were unaware of the envelope allocation sequence. Participants and outcome assessors did not know which group had been assigned to for the duration of the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet Rich Plasma (Active Comparator): In the operating room before the start of each procedure, approximately 15 cm of whole blood was drawn from the uninvolved arm of each patient in the intervention group (group I) into a 20 ml sterile syringe containing citrate for anticoagulation. The blood was immediately centrifuged at 3200 Revolutions per Minute (PRM). Following 15 minutes of centrifugation, 4 - 5 mL of PRP was obtained. Then, the PRP was buffered by using sodium bicarbonate. After closure of the fascia and prior to skin closure, PRP was directly applied to the subcutaneous tissue of the wound site by using a sterile syringe.
  Interventions: Drug: Platelet rich plasma
- control group (No Intervention): In the control group (group II), the patients did not receive topical treatment and the subcutaneous tissue was cleaned with normal saline before skin closure

INTERVENTIONS:
Drug: Platelet rich plasma — approximately 15 cm of whole blood was drawn from the uninvolved arm of each patient in the intervention group (group I) into a 20 ml sterile syringe containing citrate for anticoagulation. The blood was immediately centrifuged at 3200 Revolutions per Minute (PRM). Following 15 minutes of centrifugation, 4 - 5 mL of PRP was obtained. Then, the PRP was buffered by using sodium bicarbonate.
  Arms: Platelet Rich Plasma

SUMMARY:
Objective: To assess the effect of autologous Platelet Rich Plasma (PRP) on wound healing and pain perception in high risk women undergoing cesarean sections in a low resource setting.

Methods: This was a randomized controlled trial of 200 women who attended the outpatient clinic of Menoufia University Hospital for elective cesarean surgery. The women were randomly assigned to two groups. The intervention group received PRP after surgery, whereas the control group received the usual care. Outcomes included Redness, Edema, Ecchymosis, Discharge, Approximation (REEDA) scale, Vancouver scar scale (VSS), and the visual analog scale (VAS).

DETAILED DESCRIPTION:
The investigators conducted this randomized controlled trial from April 2018 to July 2020 at the Department of Obstetrics and Gynecology at Menoufia University Hospital, which is a large tertiary center in the Delta region in Egypt with a delivery rate of about 10000 per year. This study was approved by Menoufia university hospital ethical committee Institutional review board (198190PSGN33). The investigators obtained informed consent from all participants before initiating any study procedures. CONSORT guidelines were observed and completed.

The patients included in the study were between 20 and 40 years of age. Eligible women had one or more of the following risk factors: Body mass index (BMI) > 30 kglcm2, prior cesarean section, pregestational or gestational diabetes, hypertensive disorders of pregnancy, placenta Previa, twin pregnancy, anemia, and corticosteroid medication. Exclusion criteria were chronic pain disorders, hepatitis, thrombocytopenia, and coagulation disorders.

The investigators randomized participants in a 1:1 ratio to two equal groups containing one hundred patients each (intervention and control groups). A statistician not directly involved in the study prepared a computer generated randomization list and placed the allocation information in sequentially numbered sealed envelopes that were opened according to the attendance of the patients after signing the informed consent. The study authors were unaware of the envelope allocation sequence. Participants and outcome assessors did not know which group had been assigned to for the duration of the study.

In the operating room before the start of each procedure, approximately 15 cm of whole blood was drawn from the uninvolved arm of each patient in the intervention group (group I) into a 20 ml sterile syringe containing citrate for anticoagulation. The blood was immediately centrifuged at 3200 Revolutions per Minute (PRM). Following 15 minutes of centrifugation, 4 - 5 mL of PRP was obtained. Then, the PRP was buffered by using sodium bicarbonate. After closure of the fascia and prior to skin closure, PRP was directly applied to the subcutaneous tissue of the wound site by using a sterile syringe. In the control group (group II), the patients did not receive topical treatment and the subcutaneous tissue was cleaned with normal saline before skin closure. For all patients, the skin was closed with polyprolene 2-0 suture with a curved cutting needle. The patients were examined by the physicians who were blinded to the group allocation on day 1, and then day 7 and 6 months after the procedure.

Pain was evaluated by the visual analog scale system (VAS) which assesses changes of pain via a continuous measurement instrument that is operationally comprised of a horizontal line, anchored at each end by verbal descriptors such as no pain and the worst pain imaginable. The subject is asked to indicate a spot on the scale that best represents her degree of pain. The score is determined by measuring the distance (mm) between the no pain anchor to the point that the patient marks, providing a range of scores from 0 - 10. A higher score indicates greater pain intensity.

The primary outcome was the Redness, Edema, Ecchymosis, Discharge, Approximation (REEDA) scale for assessing the changes in wound healing. REEDA as a descriptive scale has 4 points in a categorical score that measures 5 items of healing: redness (hyperemia), edema, ecchymosis, discharge, and approximation of the wound edges (coaptation). Each item is rated on a scale of 0 to 3, and total scores may range from 0 to 15. A lower score indicates better healing.

The secondary outcomes were measured by Vancouver scar scale (VSS) and VAS. VSS use to detect changes of formation of keloids or hypertrophic scars. It assesses 4 subjective variables: vascularity, height/thickness, pliability, and pigmentation within a possible range of 0 - 14 for the total score.

The sample size was calculated by using Epi-Info program version 3.5.4 by adjusting confidence interval to 95%. With an alpha error of 5% and study power of 80% and assuming a clinically relevant reduction in REEDA and VSS scores based on results of previous studies, the invesigators estimated a total sample size of 182 women (91 for each group). This was increased to 200 women considering about 10% drop out rate. The data collected, were tabulated and analyzed by SPSS (statistical package for the social science software) statistical package version 20 (Chicago Inc., USA), the following tests were used; Quantitative data were expressed as mean and standard deviation (X ± SD) and analyzed by applying student t test. Qualitative data were analyzed by Chi Square test. P-value at 0.05 was used to determine significance regarded as non-significant P> 0.05, significant P≤ 0.05 or highly significant P≤ 0.001.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) > 30 kglcm2
* prior cesarean section
* pregestational or gestational diabetes
* hypertensive disorders of pregnancy
* placenta Previa
* twin pregnancy
* anemia
* corticosteroid medication

Exclusion Criteria

* • chronic pain disorders

  * hepatitis
  * thrombocytopenia
  * coagulation disorders

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Redness, Edema, Ecchymosis, Discharge, Approximation scale changes | day 1, day 7 and 6 months
  for assessing the changes in wound healing. REEDA as a descriptive scale has 4 points in a categorical score that measures 5 items of healing: redness (hyperemia), edema, ecchymosis, discharge, and approximation of the wound edges (coaptation). Each item is rated on a scale of 0 to 3, and total scores may range from 0 to 15. A lower score indicates better healing

SECONDARY OUTCOMES:
Vancouver scar scale changes. | day 1, day7, and 6 months
  Vancouver scar scale (VSS) use to detect changes of formation of keloids or hypertrophic scars. It assesses 4 subjective variables: vascularity, height/thickness, pliability, and pigmentation within a possible range of 0 - 14 for the total score. A lower score indicates better healing.
Visual Analog Scale changes | day 1, day7, and 6 months
  Pain was evaluated by the visual analog scale system (VAS) which assesses changes of pain via a continuous measurement instrument.The score is determined by measuring the distance (mm) between the no pain anchor to the point that the patient marks, providing a range of scores from 0 - 10. A higher score indicates greater pain intensity

CONTACTS AND LOCATIONS:
Overall Officials: Nabih Elkhouly, Principal Investigator — Faculty of medicine, Menoufia University, Egypt
Locations (1):
- Menoufia university hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No